CLINICAL TRIAL: NCT00916916
Title: Lanreotide Levels in Acromegaly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Other Study IDs: 15070
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Acromegaly
Keywords: Acromegaly; Lanreotide
MeSH Terms: conditions — Acromegaly | interventions — Blood Specimen Collection

GROUPS / COHORTS (1):
- Lanreotide: Patients taking lanreotide for the treatment of acromegaly.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — A blood draw will occur to take 10cc of blood to measure lanreotide levels.

SUMMARY:
Recently lanreotide (a somatostatin analog) has come into the US marketplace as a commercially available medication approved by the FDA for the treatment of acromegaly. Blood levels in patients getting this drug are unknown and it may be critical to know the levels in patients whose symptoms are poorly controlled.

This is a clinical study of a medical device where the following condition is met: This is research on a medical device for which an investigational device exemption application (21 CFR Part 812) is not required.

The study is exempt from IDE requirements under 21 CFR 812.2(c)(3):

The participants will be 10 CSMC patients who are taking Lanreotide for clinical purposes. After receiving an information sheet and providing verbal consent, the participants will go to their routine blood draw. At this time, they will have an additional 10 cc plasma drawn, which will be sent to Intersciences Institute in Inglewood California to have the lanreotide plasma levels measured.

The key points of this study are:

Patients will have blood drawn at the same time as they are having blood drawn for routine care to avoid unnecessary sticks.

No patient identifiers will be sent to the lab or to any investigators- all plasma tubes will be coded by ISI as a kit and these kits will be given to the physicians. In turn the physician will give the kit to the patients who wish to have their levels measured and the patient will take the kit with them to their routine blood draw. Following the drawing and processing of the blood we will request that the lab just drop the coded plasma tube (and the patient's height weight and monthly lanreotide dose) into the mail in the prepaid mailer. The only information that the investigators will receive is the patient's height, weight and monthly lanreotide dose and the plasma lanreotide level.

No more than 10 cc of blood (a couple of tablespoons) will be drawn for lanreotide measurement.

Whenever possible plasma (which would otherwise be discarded) will be used rather than freshly drawn blood.

All plasma will be assayed at ISI.

The patient will not be charged for the lanreotide assay, an investigational assay. The assay is currently investigational and does not have a "maker" at this time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Receiving lanreotide depot for treatment of acromegaly

Exclusion Criteria:

* Unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Cedars-Sinai Pituitary Center
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States